CLINICAL TRIAL: NCT06062472
Title: Effect of Lactobacillus Paracasei PS23 on Improving Aging and Muscle Loss in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chi-Chang Huang (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Chi-Chang Huang, Principal Investigator, National Taiwan Sport University
Organization: National Taiwan Sport University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 23-006-A2
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-04

CONDITIONS: Elderly; Muscle Loss; Depression; Anxiety
MeSH Terms: conditions — Muscular Atrophy; Depression; Anxiety Disorders | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Probiotics (Experimental): Probiotic capsules contain 10 billion CFU (colony forming units) of Lactobacillus paracasei, 2 caps daily use
  Interventions: Dietary Supplement: Probiotics
- Heat-Treated Probiotics (Experimental): heat-treated probiotic capsule contain 10 billion of Lactobacillus paracasei, 2 caps daily use
  Interventions: Dietary Supplement: heat-treated of Lactobacillus paracasei HT-PS23
- Placebo (Placebo Comparator): The placebo capsule contains microcrystalline cellulose, 2 caps daily use
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Lactobacillus paracasei PS23 will be used in this study
  Arms: Probiotics
Dietary Supplement: heat-treated of Lactobacillus paracasei HT-PS23 — heat-treated probiotic capsule contain 10 billion of Lactobacillus paracasei, 2 caps daily use
  Arms: Heat-Treated Probiotics
Dietary Supplement: Placebo — The placebo capsule contains microcrystalline cellulose, 2 caps daily use
  Arms: Placebo

SUMMARY:
This study refers to the supplementation of PS23 in human experiments to help the elderly maintain muscle mass, delay muscle loss, promote physical activity, and delay the occurrence of disability and debilitation in elderly people.

DETAILED DESCRIPTION:
Taiwan has become an aging society in recent years. There are important issues to attenuate aging and activate the potential capacity of elderly population. The physical function of middle-aged and older people will degenerate with age and produce age-related diseases. Common symptoms are organ function deterioration, and old age disability caused by malnutrition and muscle loss is also a common care problem. Therefore, how to prevent the complications of muscle loss is one of the important ten years of geriatric research. Although past research has been confirmed, it can improve the debilitating condition of the elderly through nutrition counseling and exercise intervention. However, there is not much in-depth discussion on how probiotics can improve muscle loss and delay symptoms in elderly people. Therefore, this study refers to the supplementation of PS23 in human experiments to help the elderly maintain muscle mass, delay muscle loss, promote physical activity, and delay the occurrence of disability and debilitation in elderly people. One hundred and twenty elderly people will be recruited and then divided into three groups with 40 people in each group: (A) placebo group, (B) PS23 probiotic group, (C) PS23-HT prebiotic group, supplemented for 12 weeks. The diet record, functional test and muscle mass will be carried out every six weeks after the start, to understand whether PS23 is effective in improving muscle loss and weakness in elderly people.

ELIGIBILITY:
Inclusion Criteria:

* age between 65 and 85 years old

Exclusion Criteria:

* Have taken antibiotics within one month or are receiving antibiotic treatment
* Have used probiotic products in powder, capsule or tablet form within two weeks (except for yogurt, yogurt, Yakut and other related foods)
* People allergic to lactic acid bacteria products
* Patients diagnosed with stroke or hypertension (systolic blood pressure greater than 139, diastolic blood pressure greater than 89)
* Exclusion of limbs and hips that have been replaced with artificial joints
* Persons with incapacity/insufficient decision-making ability
* Who has been determines that it is not suitable to participate in the research.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 119 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
muscle mass | From Baseline, 6 weeks and 12 Weeks Assessed
  Use dual-energy X-ray absorptiometry, DXA (Lunar iDXA, GE Healthcare, IL, USA) for no-entry measurement to determine muscle mass
30 seconds chair stand test | From Baseline, 6 weeks and 12 Weeks Assessed
  30 seconds chair stand test will be used as a self-test. Number of stands will be counted.
Grip strength | From Baseline, 6 weeks and 12 Weeks Assessed
  Use the armed grip machine to measure, hold each of the left and right hands three times until they are weak, and record the maximum value

SECONDARY OUTCOMES:
Generalized Anxiety Disorder 7-Item, GAD-7 | From Baseline, 6 weeks and 12 Weeks Assessed
  The GAD-7 Anxiety Questionnaire involves 7 items assessing how often participants have felt bothered by anxiety-related problems over the past two weeks. Each item is rated on a Likert scale from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0-21; where 0-4 = minimal anxiety; 5-9 = mild anxiety; 10-14 = moderate anxiety; 15-21 = severe anxiety
Geriatric Depression Scale, GDS | From Baseline, 6 weeks and 12 Weeks Assessed
  It consists of 30 questions questioning the mood in the last week. This short form consists of 15 questions questioning the mood of the patient. The answers are given according to the feelings in the last week; The answers are "yes" or "no" and 1 point is given for "yes" or "no" answers depending on the question. For the long form: Normal 0 - 10, Mild 11 - 20, Moderate to Severe 21 - 30.For the short form: Normal 0 - 4, Mild 5 - 9, Moderate to Severe 10 - 15.
Q-LES-Q | From Baseline, 6 weeks and 12 Weeks Assessed
  Participants who receive app-CBT will have greater improvement on quality of life, assessed using The Quality of Life, Enjoyment, and Satisfaction Questionnaire - Short Form (Q-LES-Q). The Q-LES-Q-SF is a self-report measure of subjective quality of life, containing Likert items ranging from 1 (Very Poor) to 5 (Very Good). Total scores are presented as a percentage of the maximum value (i.e., ranging from 0 to 100, with higher scores indicating greater quality of life).
Visual Analogue Scale for GI symptoms, VAS-GI | From Baseline, 6 weeks and 12 Weeks Assessed
  Visual Analogue Scale for GI symptoms, VAS-GI (visual analogue scale, VAS 0-10) was designed to measure the response of symptoms and well-being in patients after taking probiotics
PGI-C | From Baseline to 12 Weeks Assessed
  The PGIC is a scale participants use to rate the level of change they have experienced following treatment. The PGIC is a 7-point scale from 1 (very much better) to 7 (very much worse).
10 meter walk | From Baseline, 6 weeks and 12 Weeks Assessed
  Use a pyramid and a measuring tape to measure a distance of ten meters, and ask the subject to stand up from the chair, go around the pyramid and sit down, and record the time
fat percentage | From Baseline, 6 weeks and 12 Weeks Assessed
  Use dual-energy X-ray absorptiometry, DXA (Lunar iDXA, GE Healthcare, IL, USA) for no-entry measurement to determine fat percentage
One-leg stance test | From Baseline, 6 weeks and 12 Weeks Assessed
  To evaluate static balance ability
Get Up and Go test | From Baseline, 6 weeks and 12 Weeks Assessed
  To evaluate functional walking ability
Sit and Reach Test | From Baseline, 6 weeks and 12 Weeks Assessed
  To evaluate lower-limb strength and flexibility
Cardiorespiratory fitness | From Baseline, 6 weeks and 12 Weeks Assessed
  2-min step test to assess the functional capacity of the respiratory and cardiovascular systems
Safety assessment - AST | From Baseline, 6 weeks and 12 Weeks Assessed
  Safety is assessed function of liver and kidney such as AST (8-38 IU/L).
Safety assessment - ALT | From Baseline, 6 weeks and 12 Weeks Assessed
  Safety is assessed function of liver and kidney such as ALT (4-44 IU/L)
Safety assessment - Bun | From Baseline, 6 weeks and 12 Weeks Assessed
  Safety is assessed function of liver and kidney such as Bun (6-20 mg/dl)
Safety assessment - Creatinine | From Baseline, 6 weeks and 12 Weeks Assessed
  Safety is assessed function of liver and kidney such as Creatinine (0.6-1.3 mg/dl)
Stress assessment - difference of Testosterone level | From Baseline, 6 weeks and 12 Weeks Assessed
  To assess inflammation indicators, used commercial kit human Testosterone (Cayman, Mich, USA) and Elisa reader (PerkinElmer, Massachusetts, USA) for analysis Male 265-923 (in ng/dl) Female 15-70 (in ng/dl) for 19 years and older
Difference in Oxidative stress - blood level of HSCRP | From Baseline, 6 weeks and 12 Weeks Assessed
  To assess inflammation indicators, used commercial kit human CRP (Cayman, Mich, USA) and Elisa reader (PerkinElmer, Massachusetts, USA) for analysis
Gut microbiota | From Baseline 12 Weeks Assessed
  Collect the DNA of fecal flora to test the diversity and abundance of gut microbiota in Stool samples before and after probiotics
Level of Growth Differentiation Factor-15 | From Baseline, 6 weeks and 12 Weeks Assessed
  Level of Growth Differentiation Factor-15
Change in Insulin Sensitivity | From Baseline, 6 weeks and 12 Weeks Assessed
  Change in fasting glucose
The serum IL-6 level | From Baseline, 6 weeks and 12 Weeks Assessed
  the measurement of serum IL-6 level in blood
TNF-a determination using ELISA | From Baseline, 6 weeks and 12 Weeks Assessed
  A serum level of TNF-a was determined by quantitative sandwich enzyme immunoassay (R&D Systems, Inc., Minneapolis, MN, USA) guided by to the manufacturer's instructions. The intensity of the color was measured at 490 nm.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Sport University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided